CLINICAL TRIAL: NCT00548236
Title: Pilot Study of a Multicenter, Telephone-Based Exercise Intervention for Patients With Early-Stage Breast and Colorectal Cancer: The Active After Cancer Trial (AACT)
Brief Title: The Active After Cancer Trial (AACT)
Acronym: AACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Cancer and Leukemia Group B (Network)
Responsible Party: Principal Investigator, Jennifer A. Ligibel, MD, Assistant Professor, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 07-266
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Colorectal Cancer
Keywords: exercise intervention; AACT
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Immediate participation in a 16-week exercise program
  Interventions: Behavioral: Telephone-Based exercise intervention
- 2 (No Intervention): Control population; will receive exercise plan after 16-week control period

INTERVENTIONS:
Behavioral: Telephone-Based exercise intervention — Exercise counselling offered via telephone calls
  Arms: 1

SUMMARY:
This study is being done to determine whether a telephone-based counseling intervention can help survivors of breast and colorectal cancer increase their weekly physical activity. Observational evidence suggests that physical activity after breast and colorectal cancer diagnosis decreases recurrence rates. Unfortunately, many people become less active during cancer therapy, and a substantial proportion never return to pre-diagnosis levels of physical activity. This study looks to see if people who have recently finished chemotherapy for breast, colon or rectal cancer can be motivated to increase their exercise by talking to an exercise specialist over the phone. The study also looks at changes in mood, fatigue, fitness, fat distribution and weight.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage I-III breast or colorectal cancer
* 18 years of age or older
* Completed adjuvant treatment(for current malignancy)
* Completion of all adjuvant chemotherapy and radiation (with the exception of adjuvant herceptin and/or tamoxifen/aromatase inhibitor therapy for breast cancer patients) between 2 and 36 months prior to enrollment
* Ability to speak and read English
* Willingness to be randomized
* Medical clearance from an oncologist or primary care physician stating the participant is able to participate in an unsupervised, moderate-intensity physical activity program
* No major surgery within 2 months of study enrollment or planned during study period

Exclusion Criteria:

* Metastatic cancer
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness that would limit compliance with study requirements
* Plans to have hip or knee replacement within a year
* Participation in more than 60 minutes a week of moderate-intensity recreational activity as assessed by the International Physical Activity Questionnaire Short Form
* BMI >47

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the ability of a multi-center, telephone-based physical activity intervention to increase weekly physical activity levels in sedentary patients treated with adjuvant chemotherapy for Stage I-III breast or colorectal cancer. | months

SECONDARY OUTCOMES:
To evaluate the impact of a physical activity intervention upon fitness, exercise self-efficacy, anthropometric measures, and quality of life in a group of patients with stage I-III breast or colorectal cancer. | months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ligibel, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (9):
- United States (9):
  - University of California at San Diego, La Jolla, California
  - University of California San Francisco, San Francisco, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - New Hampshire Oncology Hematology, Concord, New Hampshire
  - Lakes Regional Healthcare Hematology Oncology, Hooksett, New Hampshire
  - Rosewell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York, East Syracuse, New York
  - Ohio State University, Columbus, Ohio
  - Vermont Cancer Center, Burlington, Vermont